CLINICAL TRIAL: NCT03877718
Title: A Study to Assess the Efficacy and Safety of Oral CL-H1T in the Treatment of Acute Migraine Pain, With or Without Aura, and the Prevention of Migraine Associated Nausea and Vomiting.
Brief Title: A Study to Assess the Efficacy and Safety of Oral CL-H1T in the Treatment of Acute Migraine Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charleston Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL02-204
Record Dates: First submitted 2019-03-05; First posted 2019-03-18 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-03

CONDITIONS: Migraine; Pain; Nausea; Vomiting; Aura
Keywords: Acute Migraine Pain; Acute Migraine Pain, With or Without Aura; Prevention of Migraine Associated Nausea and Vomiting (MANV)
MeSH Terms: conditions — Migraine Disorders; Pain; Nausea; Vomiting; Epilepsy | interventions — Sumatriptan; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1: CL-H1T (Experimental): Maximum dosage within a 24-hour period: One capsule of CL-H1T (total dose: sumatriptan succinate 90mg/promethazine hydrochloride 18.75mg)
  Interventions: Drug: Arm 1: CL-H1T
- Arm 2: CL-H1T (Experimental): Maximum dosage within a 24-hour period: One capsule of CL-H1T (total dose: sumatriptan succinate 90mg/promethazine HCl 37.5mg)
  Interventions: Drug: Arm 2: CL-H1T
- Arm 3: Sumatriptan succinate 100 mg (Experimental): Maximum dose within a 24 hour period: One capsule of sumatriptan succinate 100mg
  Interventions: Drug: Arm 3: Sumatriptan Succinate 100 mg capsule
- Arm 4: Promethazine HCl 18.75 mg (Experimental): Maximum dose within a 24 hour period: One capsule of promethazine HCl 18.75mg
  Interventions: Drug: Arm 4: Promethazine HCl 18.75 mg
- Arm 5: Promethazine HCl 37.5 mg (Experimental): Maximum dose within a 24 hour period: One capsule of promethazine HCl 37.5mg
  Interventions: Drug: Arm 5: Promethazine HCl 37.5 mg
- Arm 6: Placebo (Experimental): Maximum dose within a 24 hour period: One capsule of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Arm 1: CL-H1T — One capsule of CL-H1T (total dose: sumatriptan succinate 90mg/promethazine HCl 18.75 mg)
  Other Names: sumatriptan succinate 90mg/promethazine HCl 18.75mg
  Arms: Arm 1: CL-H1T
Drug: Arm 2: CL-H1T — One capsule of CL-H1T (total dose: sumatriptan succinate 90mg/promethazine HCl 37.5 mg)
  Other Names: sumatriptan succinate 90mg/promethazine HCl 37.5mg
  Arms: Arm 2: CL-H1T
Drug: Arm 3: Sumatriptan Succinate 100 mg capsule — One capsule of sumatriptan succinate 100 mg
  Other Names: Sumatriptan succinate 100 mg
  Arms: Arm 3: Sumatriptan succinate 100 mg
Drug: Arm 4: Promethazine HCl 18.75 mg — One capsule of promethazine HCl 18.75 mg
  Other Names: Promethazine HCl 18.75
  Arms: Arm 4: Promethazine HCl 18.75 mg
Drug: Arm 5: Promethazine HCl 37.5 mg — One capsule of promethazine HCl 37.5 mg
  Other Names: Promethazine HCl 37.5
  Arms: Arm 5: Promethazine HCl 37.5 mg
Other: Placebo — One capsule of placebo
  Arms: Arm 6: Placebo

SUMMARY:
A Study to Assess the Efficacy and Safety of Oral CL-H1T in the Treatment of Acute Migraine Pain.

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-Blind, Comparator-Controlled, Placebo-Controlled Study to Assess the Efficacy and Safety of Oral CL-H1T in the Treatment of Acute Migraine Pain, With or Without Aura, and the Prevention of Migraine-Associated Nausea and Vomiting (MANV)

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to give written informed consent and authorize the Health Insurance Portability and Accountability Act (HIPAA) prior to entering the study.
2. Men and women with episodic migraine who meet the criteria of the International Headache Society's Headache Classification Committee for migraine with or without aura.
3. Between the ages of 18 and 75 years of age, inclusive.
4. A history of episodic migraine for at least 1 year.
5. Maximal frequency of 8 migraine attacks per month; minimum frequency of 2 migraine attacks per month; at least 48 hours of headache-free time between migraine attacks.
6. Maximum total headache days of 14 per month.
7. History of migraine headache with nausea ≥ 50% of the time.
8. Able and willing to complete an electronic diary (eDiary) to record the details of a migraine attack treated with investigational treatment.
9. Able to swallow a capsule whole.
10. Report headache on the Headache Pain Scale at Baseline before treatment.
11. Report the presence of nausea on the Nausea Scale at Baseline before treatment.
12. Women of childbearing potential (WOCBP) must practice an acceptable method of birth control (acceptable methods of birth control in this study include: surgical sterilization, intrauterine device, oral contraceptive, contraceptive patch, long-acting injectable contraceptive, partner's vasectomy, or a double-barrier method [condom or diaphragm with spermicide]). Use of intrauterine devices and hormonal contraceptives must begin at least 8 weeks prior to Screening.
13. Willing and able to comply with the protocol requirements for the duration of the study.

Exclusion Criteria:

1. A clinically significant or unstable medical or surgical condition that would preclude safe and complete study participation. Such conditions may include cardiac, respiratory, hepatic, renal or metabolic diseases, peripheral vascular disease, any systemic disease, acute infection, or neurological disease (including Parkinson's Disease or other condition associated with a movement disorder), current malignancy or recent history (within 5 years) of malignancy (other than squamous cell or basal cell carcinoma) or any medical condition that, in the opinion of the Investigator, makes the subject unsuitable for participation in the study.
2. A positive saliva screen for alcohol or a positive urine drug screen for cocaine, narcotics, benzodiazepines, opioids, tetrahydrocannabinol (THC), barbiturates, amphetamines, or any prescription drugs unless such a positive result can be explained by stated concomitant medications.
3. Regularly smoke cigarettes or use opiate analgesic drugs, benzodiazepines, ergot containing drugs, alcohol, THC, or other drugs of abuse that, at the discretion of the Investigator, may interfere with the evaluation of the endpoints in the trial.
4. Unstable use of prophylactic migraine medication (eg, change of dose or type of medication) during the 30 days prior to Screening Visit.
5. Subjects using monoamine oxidase-A (MAO-A) inhibitors and who cannot be washed out.
6. Subjects using selective serotonin reuptake inhibitors (SSRIs), serotonin norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, THC, or systemic corticosteroids over the past month prior to the Screening Visit.
7. Daily use of antipsychotics at least 15 days prior to randomization.
8. Medication overuse:

   1. Opioids for headache ≥ 10 days during the 90 days prior to Screening Visit;
   2. Combination medications that contain an opioid and/or barbiturate (eg, Fiorinal®) ≥ 10 days during the 90 days prior to Screening Visit.
   3. Nonsteroidal anti-inflammatory drugs (NSAIDs) or other simple medications ˃ 14 days a month during the 90 days prior to Screening Visit.
   4. Triptans or ergots ≥ 10 days a month during the 90 days prior to Screening Visit.
9. Use of mini prophylaxis for menstrual migraine.
10. History of allergic reaction or drug sensitivity to any triptans.
11. History of allergic reaction or drug sensitivity to promethazine.
12. History of allergic reaction or drug sensitivity to acetaminophen.
13. History of extrapyramidal reaction (eg, akathisia or dystonia) to neuroleptic treatments.
14. Subjects who are pregnant (positive urine hCG: Human chorionic gonadotropin test at Screening Visit) or breastfeeding.
15. Use of experimental or investigational treatments and/or participation in drug clinical studies within the 6 months before the Screening Visit.
16. Subjects who are employees of the Sponsor.
17. Relatives of, or staff directly reporting to, the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who are pain-free 2 hours after taking investigational treatment | 2 hours
Percentage of subjects who are nausea-free 2 hours after taking investigational treatment | 2 hours

SECONDARY OUTCOMES:
Percentage of subjects with no vomiting 2 hours after taking the investigational treatment | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bernard P. Schachtel, MD, Study Chair — Charleston Laboratories
Locations (3):
- United States (3):
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Harmony Clinical Research, Inc., North Miami Beach, Florida
  - Mountain View Cl inical Research, Inc., Greer, South Carolina

IPD SHARING:
Plan to Share IPD: No